CLINICAL TRIAL: NCT05781139
Title: Comparative Study Between Alzheimer's and Multi-infarct Dementia Regarding to Clinical Aspect, Biomarker, and Cortical Excitability
Brief Title: Comparative Study Between Alzheimer's and Multi-infarct Dementia
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, AAEsraa, Assistant Lecturer, Assiut University
Other Study IDs: Dementia
Record Dates: First submitted 2023-02-20; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (4):
- Early onset Alzhiemer: before age of 65 and above age of 50
  Interventions: Diagnostic Test: levels of Neurofilaments (NfL) in serum
- Late onset Alzhiemer: Above the age of 65
  Interventions: Diagnostic Test: levels of Neurofilaments (NfL) in serum
- Vascular dementia: Any patient diagnosed with vascular dementia
  Interventions: Diagnostic Test: levels of Neurofilaments (NfL) in serum
- control group: persons who has no dementia
  Interventions: Diagnostic Test: levels of Neurofilaments (NfL) in serum

INTERVENTIONS:
Diagnostic Test: levels of Neurofilaments (NfL) in serum — the levels Neurofilaments (NfL) (Abcam, USA), C-X-C motif chemokine 13 (CXCL13) and Chitinase 3-like Protein 1 (Sigma-aldrich, Germany) will be determined in the serum and CSF (if available) in the different participant groups.

SUMMARY:
Dementia is a neurological disease that causes cognitive and behavioral impairments that could ultimately interfere with the ability to function at work or to do the usual daily activities. It is recognized as a healthcare and social burden and remains challenging in terms of proper diagnosis and treatment.

DETAILED DESCRIPTION:
Biomarkers are needed to identify at-risk individuals, stage their disease, and track disease progression. Such biomarkers should be noninvasive, inexpensive, and simple to acquire. Neurodegeneration biomarkers in CSF include neurofilament light (NfL), Chitinase 3-like protein 1 (CHI3L1). NfL for example increases in several neurologic conditions, including AD. In addition, NfL can be detected in serum using standard immunoassay formats. Higher CSF levels of CHI3L1 are seen in patients with neurological disorders such as MS patients experiencing relapses of MS. In addition, C-X-C motif chemokine 13 (CXCL13) is a crucial homeostatic chemokine expressed in lymphoid organs, and it is essential for the recruitment and compartmentalization of lymphocytes. In MS, CXCL13 regulates homing of B cells and subsets of T cells to inflammatory foci in CNS by interacting with the CXCR5 receptor. The levels of CXCL13 are elevated in the CSF of patients with MS compared to healthy controls, as well as in other neuroinflammatory diseases. CXCL13 may be considered a CSF biomarker of intrathecal B cell response, as its levels correlate with the count of B cells, the IgG index, and the presence and OCBs in the CSF.

Transcranial magnetic stimulation (TMS) assesses several cortical properties such as excitability, plasticity, and connectivity in humans. TMS has been applied to patients with dementia, enabling the identification of potential markers of the pathophysiology and predictors of cognitive decline; moreover, applied repetitively, TMS holds promise as a potential therapeutic intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women of at least 50-80 years of age.
2. Are reliable in individual data and willing to make themselves available for the duration of the study
3. Clear written informed consent obtained from 1st degree of relative from each patient participant and control himself in the trial.

Exclusion Criteria:

1. age below 50 years and above 80 years.
2. other neurological disorders or psychiatric disorders; previous history of stroke; metabolic disturbance; other major medical illnesses; epilepsy; inflammatory, autoimmune, or infectious disease; metallic objects in the body; craniotomy in the past.
3. Presence of clinically significant medical or psychiatric condition that may increase the risk associated with the study
4. Participation in any other type of medical research that may interfere with the interpretation of the study.
5. Patients with severe motor disability (bed-ridden) that may interfere with the study procedure.
6. Patients with history of seizures or epilepsy including history in a first degree relative

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: case control study, it will include 4 groups of dementia patients in early and late onset, and control healthy group matching with age, sex and educational state.
  The study will include 19 patient of each dementia type and 19 controls, each dementia patients were diagnosed according to the international classification of disease 10th revision ICD 10.
  Total score of Mini-mental state examination is <24 or 22 in Mini-mental state examination will be used as a screening test for detection of cases.
Sampling Method: Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2025-07-21 (Estimated); Study Completion 2026-02-21 (Estimated)

PRIMARY OUTCOMES:
detect difference between multiple types of dementia (Alzheimer's disease with early onset, and late-onset as well as multi-infarct dementia ) | 2 years
  detect difference between multiple types of dementia (Alzheimer's disease with early onset, and late-onset as well as multi-infarct dementia ) regarding clinical profile, biomarkers, and cortical excitability

CONTACTS AND LOCATIONS:
Overall Officials: Eman M Khedr, professor, Study Chair — Assiut University
Locations (1):
- Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antczak J, Rusin G, Slowik A. Transcranial Magnetic Stimulation as a Diagnostic and Therapeutic Tool in Various Types of Dementia. J Clin Med. 2021 Jun 28;10(13):2875. doi: 10.3390/jcm10132875. PMID 34203558
- [Background] Elshahidi MH, Elhadidi MA, Sharaqi AA, Mostafa A, Elzhery MA. Prevalence of dementia in Egypt: a systematic review. Neuropsychiatr Dis Treat. 2017 Mar 6;13:715-720. doi: 10.2147/NDT.S127605. eCollection 2017. PMID 28293113
- [Background] Weston PSJ, Poole T, Ryan NS, Nair A, Liang Y, Macpherson K, Druyeh R, Malone IB, Ahsan RL, Pemberton H, Klimova J, Mead S, Blennow K, Rossor MN, Schott JM, Zetterberg H, Fox NC. Serum neurofilament light in familial Alzheimer disease: A marker of early neurodegeneration. Neurology. 2017 Nov 21;89(21):2167-2175. doi: 10.1212/WNL.0000000000004667. Epub 2017 Oct 25. PMID 29070659